CLINICAL TRIAL: NCT03903250
Title: Effects of A-GPC on Reaction Time and Cognitive Function Under Acute Sleep-Deprived Conditions
Brief Title: Effects of A-GPC on Reaction Time and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mary Hardin-Baylor (Other)
Collaborators: Chemi Nutra, LLC. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: AGPC-1
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Cognitive Change; Reaction Time
Keywords: A-GPC; focus; non-resistance trained
MeSH Terms: interventions — Sugars

STUDY DESIGN:
Intervention Model Description: Two groups: placebo and active
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sugar (Placebo Comparator): 100% soluble in liquid. 4 oz. taken in the morning of testing sessions.
  Interventions: Dietary Supplement: Sugar
- A-GPC (Experimental): 100% soluble in liquid. 4 oz. taken in the morning of testing sessions.
  Interventions: Dietary Supplement: A-GPC

INTERVENTIONS:
Dietary Supplement: A-GPC — Taken orally in liquid form
  Arms: A-GPC
Dietary Supplement: Sugar — Taken orally in liquid form
  Arms: Sugar

SUMMARY:
This is a randomized, double blind, crossover design study which measures the effect of alpha-glycerylphosphorylcholine (A-GPC) on reaction time and cognitive function in non-resistance trained males and females. Participants will complete baseline testing and then be randomized into one of two crossover treatments. Participants will report to the lab for five consecutive days whilst only getting a maximum of five hours of sleep per night from Monday through Thursday night. Once testing is complete on Friday, participants will receive a one week washout period then return to complete the opposite treatment.

DETAILED DESCRIPTION:
Subjects expressing interest in doing the study will be interviewed in the UMHB Human Performance Lab (HPL) to determine whether they qualify to participate in the study. Upon qualification, participants will be scheduled a familiarization session in which participants will be taught how to use the Makoto Arena, a reaction time machine. Participants will then schedule their first testing session which will include: questionnaires, hemodynamic measures, reaction time testing, cognitive function testing via ImPACT, an acute exercise bout, reaction time testing, and cognitive function testing via ImPACT. Participants will then be randomized into one of two treatments.

Supplementation protocol: Participants will be randomly assigned into one of two treatments and will be given 4oz of either a placebo or active treatment mixed in orange flavored Gatorade everyday for 5 days. On Monday, participants will consume the beverage after testing is complete. Tuesday through Friday the beverage will be consumed as the participants arrive in the HPL.

On Mondays and Fridays, testing will be as follows: questionnaires, hemodynamic measures, reaction time testing, cognitive function testing via ImPACT, an acute exercise bout, reaction time testing, and cognitive function testing via ImPACT. On Tuesdays and Thursdays, participants will come check into the HPL for 30 minutes. On Wednesday, participants will come into the HPL to complete the acute exercise bout. To control their sleep to the best of our ability, participants are required to send emails every 30 minutes beginning at 10pm until their designated sleep time so the investigators know the participants are not asleep and gaining more than 5 hours of sleep.

ELIGIBILITY:
Inclusion Criteria

* Participants will be male or female between the ages of 18-35 years;
* Participants regularly sleep >7.5 hours per night;
* Participants have not been consistently resistance training for the past 6 months;
* Participant has provided written and dated informed consent to participate in the study;
* Participant is willing and able to comply with the protocol;
* Participant is apparently healthy and free from disease, as determined by a health history questionnaire;
* Participants agrees to not drive or operate heavy machinery while under sleep deprivation as a result of the study (Tuesday-Saturday);

Exclusion Criteria

* Participant currently smokes or have quit within the last 6 months;
* Participant is medically prescribed by a physician to take over the counter medications including medications related to insomnia or sleep aids (such as melatonin);
* Participant is medically diagnosed with a mental health/psychological disorder or suspected of having a mental health/diagnostic disorder that would be influenced or made worse by sleep deprivation;
* Participant is allergic to any ingredient in the nutritional supplement or placebo;
* Participant may be pregnant, is pregnant, is trying to become pregnant, or is breastfeeding;
* Participant has a major exam or academic requirement that will fall during the sleep deprived portion of the study (Tuesday-Friday)
* Participant reports any unusual adverse events associated with this study that in consultation with the study investigators or their doctor recommends removal from the study;
* Participants fail to abstain from operating motor vehicles or heavy machinery;

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
Effects of A-GPC on Reaction Time | within 5 days
  The primary purpose of this investigation is to determine the effectiveness of alpha-glycerylphosphorylcholine (A-GPC) on changes in reaction time in young, non-resistance trained males and females. This will be accomplished by observing changes in reaction time via the Makoto Arena. The Makoto Arena is an instrument that utilizes lights and noises to assess reaction time. Participants are required to hit the lights when they appear on the tower as fast as possible. Participants are instructed to hit as many lights as fast as possible to acquire a score that consists of the following: number of targets hit, number of targets that appeared, average reaction time, and percentage of targets hit.
Effects of A-GPC on Mental Alertness | within 5 days
  The primary purpose of this investigation is to determine the effectiveness of alpha-glycerylphosphorylcholine (A-GPC) on changes in mental alertness in young, non-resistance trained males and females. This will be accomplished by observing changes in ImPACT test scores before and after acute exercise, and after 4 days of sleep deprivation defined as only 5 hours of sleep per night. The ImPACT test measures cognitive function via the following tests: verbal memory, visual memory, symbol matching, color matching, and a three letter sequence memory test. For the verbal and visual memory tests, a composite score is taken between 0-100 with 100 indicating best cognitive performance and 0 indicating the worst cognitive performance. For the symbol matching and color matching, a visual motor composite score is taken from 0-60 with 60 indicating the best cognitive performance and 0 indicating the worst cognitive performance.
Effects of A-GPC on Mental Fatigue | within 5 days
  The primary purpose of this investigation is to determine the effectiveness of alpha-glycerylphosphorylcholine (A-GPC) on changes in mental fatigue in young, non-resistance trained males and females. This will be accomplished by observing changes in ImPACT test scores before and after acute exercise, and after 4 days of sleep deprivation defined as only 5 hours of sleep per night. The ImPACT test measures cognitive function via the following tests: verbal memory, visual memory, symbol matching, color matching, and a three letter sequence memory test. For the verbal and visual memory tests, a composite score is taken between 0-100 with 100 indicating best cognitive performance and 0 indicating the worst cognitive performance. For the symbol matching and color matching, a visual motor composite score is taken from 0-60 with 60 indicating the best cognitive performance and 0 indicating the worst cognitive performance.

CONTACTS AND LOCATIONS:
Overall Officials: Lemuel W Taylor IV, PhD, Principal Investigator — UMHB Human Performance Lab
Locations (1):
- UMHB Human Performance Lab, Belton, Texas, United States